CLINICAL TRIAL: NCT01148030
Title: Impact of Pre-surgical Nasal Bacterial Reduction on Postoperative Surgical Site Infections / Standard Care Change
Status: Terminated | Type: Observational
Why Stopped: Outcome measures for pre-intervention were much lower than anticipated.
Sponsor: 3M (Industry)
Collaborators: Sharp HealthCare (Other)
Responsible Party: Sponsor
Other Study IDs: 11319
Record Dates: First submitted 2010-06-18; First posted 2010-06-22 (Estimated); Last update posted 2014-03-03 (Estimated); Status verified 2014-02

CONDITIONS: Surgical Site Infection
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Single: 3M Skin and Nasal Antiseptic
  Interventions: Drug: 3M Skin and Nasal Antiseptic

INTERVENTIONS:
Drug: 3M Skin and Nasal Antiseptic — Intra-nasal dosing

SUMMARY:
Patients presenting in the Emergency Department or admitted to the hospital with displaced hip fractures who require hemiarthroplasty or open reduction internal fixation or with spinal instability/fractures in need of urgent surgical intervention will receive treatment to reduce the number of microorganisms in their nose prior to surgery. After surgery, the subjects will be observed for any surgical site infections.

DETAILED DESCRIPTION:
Infection rate study.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting in the Emergency Department or admitted to the hospital with displaced hip fractures who require hemiarthroplasty or open reduction internal fixation or with spinal instability/fractures in need of urgent surgical intervention will be enrolled in the study.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Emergent Hip Fractures
Sampling Method: Probability Sample
Enrollment: 333 (Actual)
Dates: Start 2010-06; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Surgical Site Infection | 1 year after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Sharp Memorial Hospital, San Diego, California, United States